CLINICAL TRIAL: NCT05563519
Title: Comparison of I-Prf Impregnated Collagen With L-Prf in Terms of Postoperative Complications and Wound Healing After Lower Impacted Third Molar Teeth Surgery
Brief Title: Comparison of the Efficacy of I-Prf Impregnated Collagen and L-Prf on Healing After Impacted Third Molar Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of Oral and Maxillofacial Surgery Department, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 25.12.2020/01
Record Dates: First submitted 2022-02-14; First posted 2022-10-03 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — proliferation regulatory factors, human urine; Collagen

STUDY DESIGN:
Intervention Model Description: Fifty patients were included for the randomized, prospective, split mouth and single-blind study. Two groups were formed in the study. The lower right and lower left wisdom teeth of the patients with extraction indication for lower impacted wisdom teeth were included in separate groups. In the first group (on one side of the same patients), leukocyte platelet-rich fibrin (L-PRF, 2700rpm,12 min) was obtained after lower impacted wisdom tooth surgery, applied into the socket and sutured. The other tooth of the patient was operated 5 weeks after the operation of the region included in the first group. In the second group (to the other side of the same patient), injectable platelet-rich fibrin (I-PRF, 700rpm, 3min) was obtained and 1*2 cm type 1 collagen plug (ACE RCP, Resorbable Collagen Plug, Collagen Matrix, Inc. Oakland, New Jersey) USA)) was impregnated and applied into the socket as such. It was followed for 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-PRF + collagen (Active Comparator): I-PRF will be applied with type 1 collagen to the extraction socket after the wisdom tooth operation.
  Interventions: Procedure: I-PRF with collagen
- L-PRF (Active Comparator): Only L-PRF will be applied to the extraction socket after the wisdom tooth operation
  Interventions: Procedure: L-PRF

INTERVENTIONS:
Procedure: I-PRF with collagen — The products will be applied to the sockets after tooth extractions
  Arms: I-PRF + collagen
Procedure: L-PRF — The products will be applied to the sockets after tooth extractions
  Arms: L-PRF

SUMMARY:
Impacted third molar extraction is a very common surgical intervention. Post-procedure pain causes various post-operative changes such as edema and trismus. Minimizing these changes will enable patients to overcome the post-operative process more easily. In this study, it was aimed to compare the possible effects of I-PRF (Impregnated Platelet Rich Fibrin) type 1 collagen with L-PRF (Leukocyte Platelet Rich Fibrin) on postoperative complications and wound healing after lower impacted wisdom tooth surgery. There are studies in the literature showing that very different treatment methods are used for buried twenty-year-old surgery. However, although there are studies in which intra-socket L-PRF, I-PRF, and collagen plugs are applied, there is no accepted standard for comparing the effects of L-PRF and I-PRF impregnated type-1 collagen with each other or for postoperative comfort. The aim of the study is to observe the effect of 2 different techniques on postoperative complications and possible changes in wound healing and discuss whether there is a difference and the effective one.

DETAILED DESCRIPTION:
Fifty patients were included for the randomized, prospective, split mouth and single-blind study. Two groups were formed in the study. The lower right and lower left wisdom teeth of the patients with extraction indication for lower impacted wisdom teeth were included in separate groups. In the first group (on one side of the same patients), leukocyte platelet-rich fibrin (L-PRF, 2700rpm,12 min) was obtained after lower impacted wisdom tooth surgery, applied into the socket and sutured. The other tooth of the patient was operated 5 weeks after the operation of the region included in the first group. In the second group (to the other side of the same patient), injectable platelet-rich fibrin (I-PRF, 700rpm, 3min) was obtained and 1*2 cm type 1 collagen plug (ACE RCP(Resorbable Collagen Plug), Resorbable Collagen Plug, Collagen Matrix, Inc. Oakland, New Jersey, USA) was impregnated and applied into the socket as such. It was followed for 4 weeks. Both surgical sites were sutured with 4\0 silk sutures (18mm, 3\8 sharp, 75cm black suture). It was determined randomly which material would be used first on which side.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and over,
* Patients with semi-impacted or fully impacted wisdom teeth,
* Patients without systemic disease (According to ASA(The American Society of Anesthesiologists) classification, ASA1 individuals),
* Individuals who did not use any medication in the last two weeks.

Exclusion Criteria:

* Individuals with painful temporomandibular joint disease,
* Internal irregularity and/or inflammatory joint disease with a mouth opening of less than 25 mm,
* Pregnant and lactating individuals,
* Individuals who do not come to their postoperative controls,
* Individuals using different drugs other than those recommended,
* Individuals who are allergic to the study drugs and materials.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Evaluation | Preoperative
  Blood pressure both systolic and diastolic will measured with automatic sphygmomanometer.
Blood Pressure Evaluation | Right after the surgery
  Blood pressure both systolic and diastolic will measured with automatic sphygmomanometer.
Pain Evaluation | Postoperative 2nd day
  Patients will requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Postoperative 7th day
  Patients will requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Postoperative 14th day
  Patients will requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Pain Evaluation | Postoperative 28th day
  Patients will requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Trismus Evaluation | Postoperative 2nd day
  Postoperative trismus will evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Trismus Evaluation | Postoperative 7th day
  Postoperative trismus will evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Trismus Evaluation | Postoperative 14th day
  Postoperative trismus will evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Trismus Evaluation | Postoperative 28th day
  Postoperative trismus will evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Edema Evaluation | Postoperative 2nd day
  Postoperative edema will evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, base of the nose, labial commissura, and soft tissue pogonion, tragus) which was measured with using thread and millimeter ruler.
Edema Evaluation | Postoperative 7th day
  Postoperative edema will evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, base of the nose, labial commissura, and soft tissue pogonion, tragus) which was measured with using thread and millimeter ruler.
Edema Evaluation | Postoperative 14th day
  Postoperative edema will evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, base of the nose, labial commissura, and soft tissue pogonion, tragus) which was measured with using thread and millimeter ruler.
Edema Evaluation | Postoperative 28th day
  Postoperative edema will evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, base of the nose, labial commissura, and soft tissue pogonion, tragus) which was measured with using thread and millimeter ruler.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Ciğerim, Assoc.Prof., Study Director — Van Yuzuncu Yil University, Faculty of Dentistry
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT05563519/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT05563519/ICF_001.pdf